CLINICAL TRIAL: NCT07038512
Title: Evaluation of the Hyivy Floora Pelvic Rehabilitation Vaginal Dilator in Managing Interstitial Cystitis/ Bladder Pain Syndrome and High-tone Pelvic Floor Dysfunction
Brief Title: Evaluation of Hyivy Floora in Managing Interstitial Cystitis/Bladder Pain Syndrome/High-tone Pelvic Floor Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Hyivy Health Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00130697
Record Dates: First submitted 2025-06-12; First posted 2025-06-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Interstitial Cystitis/Painful Bladder Syndrome; Interstitial Cystitis, Chronic; High Tone Pelvic Floor Dysfunction
Keywords: bladder and pelvic pain; lower urinary tract symptoms; sexual function
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: This is a prospective single-arm proof-of-concept before-after trial evaluating pain relief following a 12-week trial of the Floora Pelvic Rehabilitation Vaginal Dilator in female's with high-tone pelvic floor dysfunction and Interstitial Cystitis/Bladder Pain Syndrome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will be instructed to use the Hyivy Floora Pelvic Rehabilitation Vaginal Dilator at least three times per week for a total of 12-weeks. Each session consists of 10 minutes of heat and 10 minutes of dilation.
  Interventions: Device: Floora Pelvic Rehabilitation Vaginal Dilator

INTERVENTIONS:
Device: Floora Pelvic Rehabilitation Vaginal Dilator — The Floora Pelvic Rehabilitation Vaginal Dilator, created by Hyivy Health Inc, is a multi-therapy hand held ergonomic intravaginal wand device that is designed to be used in the comfort of the user's home. The Floora has two main therapeutic functions, controllable dilation and thermal therapy. It is the first vaginal dilator that performs auto-dilation using one or two air chambers inflated from the device surface by an internal pump, eliminating the need for reinsertion. The device is equipped with biosensors that measure the pressure from the vaginal canal which allows this device to provide a gradual and gentle stretch to the pelvic floor muscles. The thermal therapy is achieved through an electrical circuit, changing the temperature of the device in small increments. Users are able to force-stop and change the temperature and dilation settings during a session.

SUMMARY:
The purpose of this study is to test the safety and effectiveness of the Floora Pelvic Rehabilitation Vaginal Dilator in females with Interstitial Cystitis/ Bladder pain Syndrome (IC/BPS) and High-tome Pelvic Floor Dysfunction (HTPFD). After enrollment, participants will be given a Floora device and will be instructed to use the device at least three times per week for 12-weeks in the comfort of their home. Each session consists of 10 minutes of heat and 10 minutes of dilation. All participants will be required to attend 3 in-person clinic visits and there will be two follow-up phone-calls throughout the 16-week trial period.

DETAILED DESCRIPTION:
The expansion of Interstitial Cystitis (IC) to include Bladder Pain Syndrome (BPS) started in 2002 by the International Continence Society and was further expanded in 2008 to focus on the inclusion of chronic pelvic pain, pressure, and discomfort perceived to be related to the bladder. These symptoms must occur for more than 6 weeks in the absence of infection or other identifiable cause . There has been further distinction between patients who have erosive bladder lesions (Hunner lesions) and those who do not. The Floora allows women suffering from HTPFD and IC/BPS to manage their physical therapy treatment privately and comfortably in their own space, fostering a sense of control to take an active role in their healing. This self-controlled option can reduce anxiety, improve mental well-being, and increasing adherence to dilator therapy, ultimately leading to better outcomes in managing pain, thus improving quality of life for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Biological Female
* Previously established clinical diagnosis of Interstitial Cystitis/ Bladder Pain Syndrome (IC/BPS)
* Diagnosed with High-tone Pelvic Floor Dysfunction (HTPFD)
* Current pelvic pain score of 5 or greater on an 11-point Likert Scale
* Must be willing and able to insert intravaginal device
* No cognitive deficits
* Agrees not to commence any new treatments for HTPFD or IC/BPS (medical or physical therapy) during the 12-week intervention period

Exclusion Criteria:

* History of a spinal cord injury
* Currently pregnant or lactating
* Allergy to device materials
* Active vaginal infection (e.g. vulvovaginal candidiasis, trichomonas, vaginitis, bacterial vaginosis, STIs, etc.)
* Have open wounds, cuts, or open sores present in the vaginal or pelvic area
* Recent pelvic or abdominal surgery within the last 3 months
* Currently under the care of a pelvic floor physical therapist or pelvic floor physiotherapist
* History of Neurogenic bladder
* History of bladder, uterine, ovarian or vaginal cancer
* History of radiation cystitis
* Any pelvic floor/bladder Botox use within 6 months of enrollment and no future plans for Botox injections during the study period.
* Any other medical condition or clinical finding giving reasonable suspicion of a disease or condition that contraindicates the use of the Floora, at the discretion of the Investigator

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pelvic Pain Score | Baseline
  Overall pelvic pain score, measured on an 11-point Likert scale with 0 meaning no pain and 10 meaning the worst pain imaginable.
Pelvic Pain Score | Week 6
  Overall pelvic pain score, measured on an 11-point Likert scale with 0 meaning no pain and 10 meaning the worst pain imaginable.
Pelvic Pain Score | Week 12
  Overall pelvic pain score, measured on an 11-point Likert scale with 0 meaning no pain and 10 meaning the worst pain imaginable.
Pelvic Pain Score | Week 16
  Overall pelvic pain score, measured on an 11-point Likert scale with 0 meaning no pain and 10 meaning the worst pain imaginable.

SECONDARY OUTCOMES:
O'Leary-Sant Interstitial cystitis (IC) Symptom Score | Baseline, 6-weeks, 12-weeks and 16-weeks
  The O'Leary Sant Instrument has two parts: the ICSI assesses the presence and severity of common IC/BPS symptoms, and the ICPI assesses how these symptoms are perceived by the patient, or how big of a "problem" they are perceived to be. Both components consist of 4 questions, with responses to ICSI questions ranging from 0 (not at all) to 5 (almost always) and responses to ICPI questions ranging from 0 (no problem) to 4 (big problem). A total score (ICSI+ICPI) of greater than 12 strongly suggests the diagnosis of IC/BPS, with higher numerical scores indicating increased severity of disease.
Pelvic Pain, Urgency and Frequency (PUF) Questionnaire Score | Baseline, 6-weeks, 12-weeks and 16-weeks
  The PUF patient symptom scale is a validated instrument used to assess the severity of symptoms associated with pelvic pain conditions, like IC/BPS, and the degree to which these symptoms "bother" a patient. It is separated into two subsections, the symptom score and the bother score, to produce one composite score. The symptom score is comprised of seven items addressing urinary frequency, urgency, nocturia, dyspareunia, and pelvic pain. The bother score consists of four items assessing the degree to which the evaluable symptoms trouble the patient. Each question is scored from 0 (never) to 3 (always) or 1 (mild) to 3 (severe), except for two which quantify daytime frequency and nocturia separately with scores ranging from 0 to 4. A composite score between 10 and 14 indicates a strong diagnosis of IC/BPS with higher scores reflecting a greater degree of severity of symptoms and disease progression as well as impact on quality of life.
Pelvic Floor Impact Questionnaire- Short Form 7 (PFIQ-7) | Baseline, 6-weeks, 12-weeks and 16-weeks
  The PFIQ-7 is a shortened version of the Pelvic Floor Impact Questionnaire (PFIQ). It is a health-related quality of life questionnaire for women with pelvic floor conditions. It consists of seven questions that need to answered three times each, and assesses symptoms related to the bladder/urine, vagina/pelvis, and bowel/rectum and their effect on function, social health, and mental health in the past 3 months. The responses for each question range from 0 (not at all) to 3 (quite a bit). To get scale scores, the mean of each of the three scales is individually calculated, which ranges from 0-3, this number is then multiplied by 100 and divided by 3. The scale scores are then added together to get the total PFIQ-7 score, which ranges from 0-300. A lower score indicates a lesser effect on quality of life.
The Female Sexual Functioning Index (FSFI) | Baseline, 6-weeks, 12-weeks and 16-weeks.
  The FSFI is a 19-item multidimensional self-reporting measure that quantifies female sexual dysfunction in six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Scores for the arousal, lubrication, orgasm, and pain domains range from 0 to 6 using Likert-type scales. Scores for desire range from 1.2 to 6.0, and those for satisfaction range from 0.8 to 6.0. The total score is the sum of the domain scores and ranges from 2 to 36, and the recall period is the past 4 weeks. Higher scores indicate a better level of sexual function.
The Global Response Assessment (GRA) | 12-weeks
  The GRA will be performed post-treatment to evaluate how ultimately effective this treatment is from the perspective of the participants. It is structed on a 7-point Likert scale centered at 0, indicating no change. The question is asked as follows: "As compared to when you started the current study, how would you rate your overall symptoms now?". Participants will rate their symptoms as: Markedly worse, Moderately worse Slightly worse, The same, Slightly improved, moderately improved and markedly improved.

OTHER OUTCOMES:
Hyivy Device Satisfaction Questionnaire | 12-weeks
  The Hyivy Device Satisfaction questionnaire was created by Hyivy Health Inc to gather feedback from users. It assesses the user's overall opinion of the devices usability, functionality, performance and how well it meets their needs.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Walker, PhD, Principal Investigator — Wake Forest Institute for Regenerative Medicine
Locations (1):
- Atrium Health Wake Forest Baptist Urology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hyivy Health Inc Website — https://hyivy.com/